CLINICAL TRIAL: NCT06301152
Title: Comparison of High Intensive Laser Therapy and Extracorporeal Shock Wave Therapy in Treatment of Lateral Epicondylitis: A Randomized Controlled Study
Brief Title: Lateral Epicondylitis Treatment High Intensive Laser Therapy and Extracorporeal Shock Wave Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-22-1905
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; High Intensive Laser Therapy; Extracorporeal Shock Wave Therapy; Musculoskeletal ultrasound
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: two different treatment modalities were applied in two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensive laser (Experimental): high-intensity laser was applied 3 times in a week, for three weeks, total of 9 sessions
  Interventions: Device: high intensive laser
- extracorporeal shock wave therapy (Experimental): extracorporeal shock wave therapy was applied once a week, for three weeks total of 3 sessions
  Interventions: Device: extracorporeal shock wave therapy

INTERVENTIONS:
Device: high intensive laser — high-intensity laser ,three times in a week, for three weeks, 9 session
  Arms: high intensive laser
Device: extracorporeal shock wave therapy — extracorporeal shock wave therapy, once a week, for three weeks ,3 times,
  Arms: extracorporeal shock wave therapy

SUMMARY:
Objectives: This study aims to evaluate and compare the short-term efficacy of high-intensity laser therapy (HILT) and extra corporeal shock wave therapy(ESWT) on pain, sensitivity, handgrip strength, and functions in the treatment of lateral epicondylitis (LE).

Material and methods: Forty five participants (age range, 18 to 65 years) with unilateral elbow pain were randomized into two groups. HILT group (n = 22) and the ESWT group (n = 23). The HILT and ESWT were administered three times a week for three weeks, and each treatment was combined with exercises. All patients in both groups were evaluated with ultrasonography for common extensor tendon(CET) thickness. A visual analog scale (VAS), Quick Disabilities of the Arm, Shoulder, and Hand (QDASH), and hand grip strength test were used to evaluate the patients before, one, and six weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Lateral epicondylitis
* Age >18

Exclusion Criteria:

* Operation history about elbow
* Received physical therapy, or had a steroid injection to the elbow in the three months
* Cervical radiculopathy,
* Elbow deformities,
* Fibromyalgia syndrome,
* Carpal tunnel syndrome,
* Neurological impairments in the upper extremity,
* Chronic inflammatory conditions,
* Hemophilia,
* Pregnant,
* History of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Baseline, 1 week and 6 weeks
  score 0-10, 0 minimum value, mean is no pain, score 10 is maximum value, pain is very severe

SECONDARY OUTCOMES:
Quick Disability Arm, Shoulder and Hand questionary, | Baseline, 1 week and 6 weeks
  Quick Disability Arm, Shoulder and Hand questionary, minimum score 0 maximum score 100, high score value is associated with poor functional status
hand grip strength | Baseline, 1 week and 6 weeks
  evaluates the maximum isometric contraction strength of hand and forearm muscles, 20-69 age male 47-40kg, female 30-24kg is normal value. ow value is associated with poor function
musculoskeletal ultrasonography | Baseline, 1 week and 6 weeks
  common extensor tendon thickness;>0.40-0.41cm measurement result is associated with thickening of the tendon

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Esra Bilir, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No